

# **Statistical Analysis Plan**

PROTOCOL AEGR-734-401 (V4.0, 08FEB2018)

A 36-MONTH, MULTICENTER, OPEN LABEL PHASE 4 STUDY TO EVALUATE THE IMMUNOGENICITY OF DAILY SC METRELEPTIN TREATMENT IN PATIENTS WITH GENERALIZED LIPODYSTROPHY

**SPONSOR:** AMRYT PHARMACEUTICALS

**AUTHOR:** TRACY FRANKLIN, TINGXUAN LI, IMAANI EASTHAUSEN, LEONOR

**RODRIGUES** 

VERSION NUMBER AND DATE: V2.1, 13MAR2024

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy

Author: Tracy Franklin, Tingxuan Li, Imaani Easthausen, Leonor Rodrigues Version Number: 2.1



Statistical Analysis Plan Template

## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan (V2.1, 13MAR2024) for Protocol AEGR-734-401 (V4.0, 08FEB2018).

The SAP signature page applies to both SAP text and SAP Templates (outputs shells or Tables/Listings/Figures (TLFs) shells). Templates must be sent to the customer with the first draft SAP text.

| | Name | Signature | Date |
|---|---|---|---|
| Author: | Imaani Easthausen | DocuSigned by: Imaani Earthauren | 13-Mar-2024 |
| Position: | Senior Biostatistician | C8854A1FE2E8486 | |
| Company: | IQVIA | 33334711 E2E0430 | |

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Janet Boylan | Docusigned by: Janut Boylan ASE2CSEA84644FC | 28-Mar-2024 |
| Position: | Head of Clinical Operations | | |
| Company: | Amryt Pharma DAC | | |
| Approved By: | Brian Mangal | DocuSigned by: Brian Mangal FA68091E7FAE42C | 20-Mar-2024 |
| Position: | Contract Statistician | | |
| Company: | Amryt Pharma DAC | | |
| Approved By: | Orla Casey | DocuSigned by: ONA CASLY 957E4F8B479F407 | 19-Mar-2024 |
| Position: | Translational and Immunogenicity Lead | | |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Version Date: 13MAR2024

Copyright © 2018 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




#### Statistical Analysis Plan

| Company: | Amryt Pharma DAC |
|----------|------------------|

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




# **MODIFICATION HISTORY**

| Unique | Date of the Document Version | Author | Significant Changes from |
|---|---|---|---|
| Identifier | | | Previous Authorized Version |
| for this | | | |
| Version | | | |
| 1.0 | 02AUG2019 | Tracy | Not Applicable – First version |
| | | Franklin | |
| 2.0 | 09FEB2024 | Tracy | Study Objectives: Added exploratory |
| | | Franklin, | objectives |
| | | Tingxuan Li, | Planned Analyses: Added discussion of dry |
| | | Imaani | run |
| | | Easthausen, | Analysis Sets: |
| | | Leonor | <ul> <li>Added clarification that EAS varies</li> </ul> |
| | | Rodrigues | by both measure of interest and |
| | | | timepoint |
| | | | <ul> <li>Clairfied that EAS will be used in</li> </ul> |
| | | | primary and effectiveness analyses |
| | | | General Considerations: |
| | | | <ul> <li>Updated software versions</li> </ul> |
| | | | <ul> <li>Added discussion of when partial</li> </ul> |
| | | | date imputations are applicable |
| | | | Output Presentations: Added discussion of |
| | | | additional data visualizations to be generated |
| | | | as needed and/or appropriate |
| | | | Dispositions and Withdrawals: |
| | | | Added analyses for patients |
| | | | receiving at least one dose of |
| | | | Metreleptin, patients valid for the |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




| EAS, and total study participation in |
|---------------------------------------------------|
| years |
| Demographic and Other Baseline |
| Characteristics: Added derivation for age at |
| informed consent |
| Medical History: |
| <ul> <li>Updated definition of medical</li> </ul> |
| history to align with the CRF. |
| <ul> <li>Added derivation for age at</li> </ul> |
| lipodystrophy diagnosis |
| Study Medicaiton Exposure: Updated |
| derivation for duration of exposure |
| accounting for interruptions |
| Primary Immunogenicity Analysis: |
| o Added analysis set for the primary |
| analysis |
| o Added descriptions of the primary |
| analyses to be performed |
| o Added all relevant derivations for |
| primary analyses |
| Exploratory Analyses: Added fasting plasma |
| glucose and leptin/metreleptin concentration |
| as exploratory variables |
| Safety Outcomes: |
| o Added definitions of AESIs |
| o Added logic for selection of events |
| to include in AE tables stratified by |
| immunogenicity variables |
| Updated data windowing conventions |
| Updated partial date conventions |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy





#### Statistical Analysis Plan

| | | | • | Overall improvement of document structure, language and consistency |
|---|---|---|---|---|
| 2.1 | 13MAR2024 | Imaani | • | Windowing conventions updated. There was |
| | | Easthausen, | | an issue with some of the scheduled days. |
| | | Leonor | | Now all of them are calculated as follows: |
| | | Rodrigues | | floor (Study Month Number * 30.4). |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




# TABLE OF CONTENTS

| 1. | | REVIATIONS | | |
|---|---|---|---|---|
| 2. | | ODUCTION | | |
| <b>3.</b> | | DY OBJECTIVES | | |
| | 3.1 | Primary Objectives | | |
| | 3.2 | Secondary Objectives | | |
| | 3.3 | Safety Objectives | | |
| | 3.4 | Exploratory Objective | | |
| 4. | | DY DESIGN | | |
| | 4.1 | General Description | | |
| | | Figure 1: Study Schematic | | 12 |
| | 4.2 | Schedule of Events | | |
| | 4.3 | Changes to Analysis from Protocol | | |
| <b>5.</b> | <b>PLA</b> | NNED ANALYSES | •••••• | 12 |
| | 5.1 | Final Analysis | | |
| <b>6.</b> | ANA | LYSIS SETS | •••••• | 13 |
| | 6.1 | Full Analysis Set (FAS) | | 13 |
| | 6.2 | Safety Analysis Set (SAF) | | |
| | 6.3 | Effectiveness Analysis Set (EAS) | | 13 |
| <b>7.</b> | GENERAL CONSIDERATIONS | | | |
| | 7.1 | Baseline | | 13 |
| | 7.2 | Software Version | | 13 |
| <b>8.</b> | STAT | FISTICAL CONSIDERATIONS | ••••• | 14 |
| | 8.1 | Statistical Summaries, Tests and Confidence Interva | ls | 14 |
| | 8.2 | Missing data | | 14 |
| 9. | OUT | PUT PRESENTATIONS | ••••• | 14 |
| <b>10.</b> | DISP | OSITION AND DISCONTINUATIONS | ••••• | 14 |
| | 10.1 | Derivations | | 15 |
| 11. | <b>DEM</b> | OGRAPHIC AND OTHER CHARACTERISTICS | | 15 |
| | 11.1 | Derivations | | 15 |
| <b>12.</b> | MED | ICAL HISTORY CONDITIONS AND SURGERIA | ES | 15 |
| | 12.1 | Derivations | | 16 |
| 13. | MED | ICATIONS | | 16 |
| 14. | | OY MEDICATION EXPOSURE | | |
| | 14.1 | Derivations | | |
| Doc | ument: | Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, G | Open Label Phase 4 Study | to Evaluate the |
| | | Immunogenicity of Daily SC Metreleptin Treatment in Patients with | Generalized Lipodystropl | ny |
| Auth | nor: | Tracy Franklin, Tingxuan Li, Imaani Easthausen, Leonor Rodrigues | Version Number: | 2 |
| | | | Version Date: | 13MAR202 |



| 15 | PRIN | ARY ANALYSIS – IMMUNOGENICITY | 17 |
|---|---|---|---|
| 10. | | Primary Analysis Variables | |
| | | Primary Analysis Description, Derivations, and Definitions | |
| 16. | | ONDARY ANALYSIS – IMMUNOGENICITY | |
| 17. | | ETY OUTCOMES. | |
| L / • | 17.1 | | |
| | - / | Physical Examination. | |
| | | Vital Signs | |
| | 17.5 | 17.3.1 Derivations | |
| | 174 | Laboratory Evaluations | |
| 18. | | LORATORY ANALYSES – EFFECTIVENESS | |
| 10. | | Exploratory Analysis Variables | |
| | | Exploratory Analysis Description, Derivations, and Definitions | |
| 19. | | ENDIX 1. PARTIAL DATE CONVENTIONS | |
| | | ENDIX 1. TARTIAL DATE CONVENTIONS | |
| <b>∠</b> ∪• | $\Delta III$ | ייייייייייייייייייייייייייייייייייייי | |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




### 1. ABBREVIATIONS

| ADA | Anti-drug antibody |
|---------|-----------------------------------------------|
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ATC | Anatomic therapeutic class |
| BMI | Body mass index |
| CI | Confidence interval |
| CRF | Case report form |
| DILI | Drug induced liver injury |
| EAS | Effectiveness analysis set |
| ECLIA | Electrochemiluminescence immunoassay |
| FAS | Full analysis set |
| HbA1c | Hemoglobin A1c |
| HuL | Human leptin |
| MEASuRE | Metreletpin Effectiveness and Safety Registry |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRD | Minimum required dilution |
| NAb | Neutralizing antibodies |
| PT | Preferred term |
| RB | Receptor blocking |
| RWES | Real-world evidence solutions |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SC | Subcutaneous |
| SOC | System organ class |
| TEAE | Treatment emergent adverse event |
| TLFs | Tables, listings and figures |
| WHO-DD | World Health Organization Drug Dictionary |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Statistical Analysis Plan

#### 2. INTRODUCTION

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of the effectiveness and safety data for Protocol AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Immunogenicity of Daily Subcutaneous (SC) Metreleptin Treatment in Patients with Generalized Lipodystrophy. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This SAP is based on the protocol number AEGR-734-401 V4.0, dated 08FEB2018 and case report forms (CRFs) V7.0, dated 28MAY2021. If there are differences between the statistical methods documented in the protocol and this document, the methods in this document will supersede what is in the protocol. Any changes from the planned analyses of the final SAP will be documented in the case study report.

#### 3. STUDY OBJECTIVES

### 3.1 Primary Objectives

The primary objective is to evaluate the immunogenicity associated with daily SC metreleptin treatment in patients with congenital or acquired generalized lipodystrophy.

### 3.2 Secondary Objectives

The secondary objective is to assess 2 methods of measuring in vitro neutralizing activity to metreleptin.

#### 3.3 Safety Objectives

The safety objectives are:

- To evaluate the safety and tolerability in relation to the development of or absence of antimetreleptin or anti-human leptin (HuL) antibodies, and/or *in vitro* neutralizing activity to metreleptin in patients with congenital or acquired generalized lipodystrophy.
- To measure *in vitro* neutralizing activity in all patients with suspected loss of response (worsening of metabolic control) or endogenous leptin action (severe infections or sepsis) at time of adverse event report.

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Statistical Analysis Plan

## 3.4 Exploratory Objective

The exploratory objective is to evaluate the efficacy achieved with daily SC metreleptin treatment in patients with congenital or acquired generalized lipodystrophy.

#### 4. STUDY DESIGN

### 4.1 General Description

This study is an open-label, Phase 4 trial to provide an assessment of the immunogenicity associated with metreleptin and of any major potential risks due to development of antibodies to metreleptin. The study is being conducted to comply with an Food and Drug Administration post-marketing requirement.

Patients who have been prescribed metreleptin for generalized lipodystrophy, who meet all enrollment criteria and who have signed informed consent for this study at Screening (Visit 1) will receive the first dose of metreleptin at Enrollment/Baseline (Visit 2) at the study site. Patients will return to the study site for follow-up and collection of blood samples at regular intervals (at Month 1, 2, 4, 6, 9, 12, 18, 24, 30, and 36), for a total of 12 visits over approximately 3 years (36 months). Eleven patients who have been prescribed metreleptin will be enrolled.

All patients, including those with suspected loss of metreleptin efficacy (worsening of metabolic control) or endogenous leptin action (serious or severe infections or sepsis) should be tested for *in vitro* neutralizing activity.

The study flow diagram is presented in **Figure 1**.

Patients who sign informed consent and meet all inclusion/exclusion criteria will be enrolled in the study. Assessments will be made at the times specified in the Study Plan (**Table 1** of protocol). At the end of the 3-year study period, patients who still have *in vitro* neutralizing activity should enroll in the separate Immunogenicity Follow-up Program for continued immunogenicity monitoring.

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




**Figure 1: Study Schematic** 



#### 4.2 Schedule of Events

The schedule of events can be found in **Table 1** of the protocol.

### 4.3 Changes to Analysis from Protocol

There are no changes to the analysis from the protocol.

### 5. PLANNED ANALYSES

The following analyses are planned for this study: 1) Final Analysis to be completed after database lock with 2) a dry run to be completed prior to database lock. The purpose of the dry run is to generate all analyses prior to database lock to ensure the planned analyses as described are appropriate. The dry run will use real study data. The results will not be shared with study sites. Any changes to the planned analyses based on the dry run will be documented in this SAP for

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




transparency. Given the key study endpoints are objective measures, the risk of bias as a result of the dry run is minimal.

#### 5.1 **Final Analysis**

All final, planned analyses identified in this SAP will be performed by IOVIA Real-World Evidence Solutions (RWES) Biostatistics following Sponsor Authorization of this SAP, Database Lock, and Sponsor Authorization of Analysis Sets.

#### 6. ANALYSIS SETS

#### 6.1 **Full Analysis Set (FAS)**

The full analysis set (FAS) will contain all enrolled subjects.

#### 6.2 Safety Analysis Set (SAF)

The safety analysis set (SAF) will contain all enrolled subjects who receive at least one documented dose of metreleptin and will be used in the assessment of safety.

#### 6.3 **Effectiveness Analysis Set (EAS)**

The effectiveness analysis set (EAS) will contain all enrolled subjects who received at least one documented dose of metreleptin and who have baseline and post-dose laboratory results on the measure of interest at the time point of interest. By definition, the EAS will vary by both measure and timepoint. The effectiveness analysis sets will be used in the primary and exploratory analyses.

#### 7. **GENERAL CONSIDERATIONS**

#### 7.1 **Baseline**

The Enrollment/Baseline Visit (Visit 2) is the baseline visit, and will be conducted within 28 days of the Screening Visit. First dose of metreleptin will be administered at Baseline after all procedures for the Screening Visit, specified in **Table 1** of the protocol, are conducted.

#### 7.2 **Software Version**

All analyses and datasets will be programmed using Statistical Analysis Software Version 9.4 or higher. R Version 4.1.3 or higher may be used to generate data visualizations as needed.

Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Document: Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy Author: Tracy Franklin, Tingxuan Li, Imaani Easthausen, Leonor Rodrigues Version Number: 2.1


Statistical Analysis Plan

#### 8. STATISTICAL CONSIDERATIONS

### 8.1 Statistical Summaries, Tests and Confidence Intervals

There will be no hypothesis testing. All data will be summarized by descriptive statistics and/or listings. Number of patients with missing data will be reported where applicable. Continuous variables will be summarized by mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized by frequency counts and percentages of each category. Missing values will be excluded from percentage calculations. Where appropriate, two-sided, 90% and 80% Clopper-Pearson exact confidence intervals (CIs) will be included as well.

## 8.2 Missing data

Generally, missing data will not be imputed. As applicable, partial dates may be imputed for the purposes of categorizing medications as prior/concomitant and defining treatment emergent adverse events (TEAEs). Partial date handling is described in **Appendix 1**. Imputed dates will NOT be presented in listings. Where applicable, counts of missing observations will be reported.

#### 9. OUTPUT PRESENTATIONS

The shell document provided with this SAP describes the presentations for this study and therefore the format and content of the summary tables, listings and figures (TLFs) to be provided by IQVIA RWES Biostatistics.

In addition to the below described analyses, other data visualizations may be generated as needed to further evaluate variables and endpoints of interest. All additional data visualizations generated will be included in the TLFs.

### 10. DISPOSITION AND DISCONTINUATIONS

Subject disposition and discontinuations will be presented for all enrolled patients (FAS). The following will be summarized: patients screened (FAS), patients receiving at least one dose of Metreleptin (SAF), patients valid for the EAS, patients completing the study, discontinuations, reasons for discontinuation, and total study participation in years. See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Statistical Analysis Plan

#### 10.1 Derivations

 Study participation duration (years) = [(end of study date – informed consent date + 1)/365.25].

#### 11. DEMOGRAPHIC AND OTHER CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the SAF. The following demographic and other baseline characteristics will be reported for this study. See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

- Age at informed consent (years)
- Sex
- Ethnicity
- Race
- Participation in Metreleptin Effectiveness and Safety Registry (MEASuRE)

Note: MEASuRE a sister study by the same Sponsor designed to evaluate the long-term safety and effectiveness of metreleptin under normal conditions of clinical practice.

#### 11.1 Derivations

• Age at informed consent (years) = [(date of informed consent signature – date of birth + 1) / 365.25].

#### 12. MEDICAL HISTORY CONDITIONS AND SURGERIES

Medical History information will be presented for the SAF. Medical History conditions and surgeries are captured in the "Medical History" CRF. Conditions will be presented based on CRF categories. Medical History captured as "Other, specify" on the CRF will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at time of locked database and presented in terms of system organ class (SOC) and preferred term (PT).

Additional details about lipodystrophy diagnosis will also be summarized:

- Age at lipodystrophy diagnosis
- Lipodystrophy subtype

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

#### 12.1 Derivations

• Age at lipodystrophy diagnosis (years) = [(date of lipodystrophy diagnosis - date of birth + 1) / 365.25].

#### 13. MEDICATIONS

Medications will be presented for the SAF and coded using the latest version of the World Health Organization Drug Dictionary (WHO-DD) at database lock. Medications will be categorized as prior or concomitant, and the total number of patients in each category will be summarized by anatomic therapeutic class level 3 and preferred name.

If it is unclear whether or not a medication is prior or concomitant due to partial dates, the worst case will be assumed (i.e., concomitant). See **Appendix 1** for handling of partial dates.

- 'Prior' medications are medications which the patient started and stopped prior to the first dose of study medication.
- 'Concomitant' medications are medications which:
  - O Started prior to, on or after the first dose of study medication and started no later than 14 days following end of study medication,
  - AND ended on or after the date of first dose of study medication or were ongoing at the end of the study.

See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

#### 14. STUDY MEDICATION EXPOSURE

The summary of study drug exposure and compliance will be based on the SAF population. According to the protocol, patients should be encouraged to continue in the study and attend all protocol-specified visits until the end of the 3-year study period, even if discontinued from metreleptin, to enable continued evaluation of immunogenicity. Patients who discontinue metreleptin may restart treatment at any time during the 3-year study period. Therefore, duration of exposure will be presented in two ways: 1) total duration of exposure, and 2) duration of exposure accounting for interruptions.

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Version Date: 13MAR2024

Copyright © 2018 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



The following will also be summarized: dose interruptions, dose reductions, and overdoses, as appropriate. An overdose is defined as a dose of metreleptin that exceeds the maximum dose of 10 mg/day for patients >40 kg (refer to the United States prescribing information) and is recorded in the CRF.

See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

#### 14.1 Derivations

- Total duration of exposure (days) = date of last study medication administration date of first study medication administration + 1.
- Duration of exposure accounting for interruptions (days) = total duration cumulative time off medication
  - Cumulative time off medication is the sum of time off medication over all medication interruptions.
  - $\circ$  Time off medication (days) = restart date stop date 1.

#### 15. PRIMARY ANALYSIS – IMMUNOGENICITY

The primary immunogenicity analysis will be performed among the EAS. Analyses will be performed as described below. Additional data visualizations may be generated as needed.

#### 15.1 Primary Analysis Variables

The primary objective is to evaluate the immunogenicity associated with daily SC metreleptin treatment in patients with congenital or acquired generalized lipodystrophy. Immunogenicity will be described using the following variables:

- Anti-metreleptin/anti-HuL binding antibody measured by anti-drug antibody (ADA) titer
- Among ADA binding positive samples:
  - o Category of *in vitro* neutralizing antibody (NAb) activity to metreleptin measured by cell-based assay titer
  - Receptor blocking\* (RB) activity measured by electrochemiluminescence immunoassay (ECLIA)
    - Titer (dilution factor)
    - Percent inhibition at minimum required dilution (MRD)

\*Referred to in the protocol as receptor binding

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Statistical Analysis Plan

### 15.2 Primary Analysis Description, Derivations, and Definitions

The presence of anti-drug antibodies will be screened using an ADA binding assay, which detects antibodies to both Metreleptin and HuL, and reported as follows:

- Positive/negative for ADA binding by study visit. Positive ADA is defined as ADA binding detected at MRD (1:10 dilution factor). Both 90% and 80% two-sided Clopper-Pearson exact CIs will be presented.
- ADA binding by study visit and titer (negative [no ADA binding detected at MRD], 1:10, 1:50, 1:250, 1:1250, 1:6250, 1:31250). Dilution factors greater than 1:31250 will not be examined.
- Ever ADA positive and time to ADA positivity. Time to ADA positive result (months) = [((date of first ADA positive result date of baseline visit) + 1)/30.4].
- Peak ADA (defined as the measurement which detects ADA binding activity at the largest dilution factor) and time to peak ADA. Time to peak ADA (months) = [((date of peak ADA date of baseline visit) + 1)/30.4].

In vitro NAb activity will be measured in a cell-based assay and categorized into A, B, C, D and E categories based on titer. Categorization will be performed by IQVIA Data Management and the resulting derived data will be provided to IQVIA RWE Biostatistics. Positive/negative for NAb activity, high positive NAb activity, and NAb titer categories will be presented by study visit along with two-sided 90% and 80% Clopper-Pearson exact CIs. The titer categories are defined as follows:

- If no activity is detected upon initial testing (1:80 dilution factor) with the cell-based assay, the result is reported as category A.
- If activity is detected at the initial test concentration, the sample is retested at the same concentration (1:80 dilution factor). If no activity is detected on retest, the initial result is attributed to assay noise, and the sample is reported as category B.
- If activity is detected on both tests at MRD, the sample is diluted and retested until activity is no longer detected. Depending on the number of dilutions required to dilute NAb activity below the detectable threshold, the result is reported as follows:
  - o If no activity is detected at 1:800 dilution factor, then category C
  - o If no activity is detected at 1:8000 dilution factor, then category D
  - o If activity is detected at 1:8000 dilution factor, then category E. Dilution factors greater than 1:8000 will not be examined.

Positive NAb activity will be defined as a titer category C, D, or E result. High positive NAb activity will be defined as a a titer category D or E result. Category D and E results are considered to represent

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




high potency NAb activity. The clinical relevance of NAb activity results in any category has not been determined, and is a topic of current investigation. The following information will be summarized:

- Ever NAb positive and time to NAb positivity. Time to NAb positivity (months) = [((date of first NAb positive result date of baseline visit) + 1)/30.4].
- Ever high NAb positive and time to high NAb positivity. Time to high NAb positivity (months) = [((date of first hight NAb positive result date of baseline visit) + 1)/30.4].
- Peak NAb (defined as the measurement which detects NAb activity at the largest dilution factor) and time to peak NAb. Time to peak NAb activity (months) = [((date of peak NAb date of baseline visit) + 1)/30.4].

RB activity of anti-metreleptin/anti-HuL will be assessed by ECLIA receptor blocking assay and reported as follows:

- Positive/negative for RB activity by study visit. Positive RB activity is defined as RB activity detected at MRD (1:6 dilution factor). Both 90% and 80% two-sided Exact CIs will be presented.
- RB activity by study visit and titer (negative [no RB activity detected at MRD], 1:6, 1:30, 1:300, 1:3000). Dilution factors greater than 1:3000 will not be examined.
- Percent inhibition at MRD by study visit
- Ever RB positive and time to RB positivity. Time to RB positivity (months) =  $[((date \ of \ first \ RB \ positive \ result date \ of \ baseline \ visit) + 1)/30.4].$
- Peak RB (defined as the measurement which detects RB activity at the largest dilution factor) and time to peak RB. Time to peak RB result (months) = [((date of peak RB date of baseline visit) + 1)/30.4].

See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

### 16. SECONDARY ANALYSIS – IMMUNOGENICITY

The secondary objective of this study is to assess 2 methods of measuring *in vitro* neutralizing activity to metreleptin:

- 1. Cell-based assay
- 2. ECLIA receptor blocking assay

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




*In vitro* neutralizing activity as measured by cell-based and ECLIA receptor blocking assays are fully described by the primary analysis (**Section 15.** Primary Analysis – Immunogenicity). There will be no formal comparison of the two assay methods. No further analyses are required to achieve the secondary objective. Additional data visualizations may be generated as needed.

#### 17. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the SAF.

#### 17.1 Adverse Events

Adverse Events (AEs) will be coded using the latest version of MedDRA, and summarized by SOC, preferred name, and intensity. Intensity is captured in the CRF. See **Section 8.1** Statistical Tests and Confidence Intervals for a description of summaries to be reported.

Adverse Events of Special Interest (AESIs) are defined as:

- The presence of Category D or E *in vitro* cell-based NAb activity (or the relevant corresponding test result from the ligand-binding method) to metreleptin
- Necrotizing pancreatitis
- Hepatic adverse events including potential drug induced liver injury (DILI)
- Severe hypoglycemia
- Severe hypersensitivity reactions
- New diagnoses of autoimmune disorders (for instance, autoimmune hepatitis, glomerulonephritis, lupus erythematosus, antiphospholipid antibody syndrome, rheumatoid arthritis)
- Autoimmune disease exacerbation
- Serious infection resulting in hospitalization
- All cancers (excluding non-melanoma skin cancer) by cancer type
- Exposed pregnancies and pregnancy outcomes.

TEAEs are defined as AEs that started or worsened in severity on or after the first dose of study medication. If it is unclear whether or not an AE is a TEAE due to partial dates, the worst case will be assumed (i.e., TEAE). See **Appendix 1** for handling of partial dates.

AEs, serious AEs (SAEs), AEs of special interest (AESIs), TEAEs, AEs possibly caused by metreleptin, and AEs leading to metreleptin discontinuation will be summarized by ADA positivity and titer, cell-based NAb positivity and titer, and RB positivity, titer, and quintile of percent

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




inhibition. For each patient, only one event of each type will be selected to include in summary outputs. If a patient has multiple events the same type, the event with the highest severity level is selected. For patients with multiple events of the same type and severity, the event corresponding to the highest titer or percent inhibition level is selected. The corresponding titer and percent inhibition level are defined by the most recent measurement occurring prior to the event start date.

See **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported. Additional data visualizations may be generated as needed.

### 17.2 Physical Examination

Physical examination will be summarized by visit. The following information will be reported (see **Section 8.1** Statistical Tests and Confidence Intervals for a description of summaries to be reported):

- General Appearance (normal, abnormal, not done)
- Respiratory (normal, abnormal, not done)
- Cardiovascular (normal, abnormal, not done)
- Abdomen (normal, abnormal, not done)
- Skin (normal, abnormal, not done)
- Head and Neck (normal, abnormal, not done)
- Lymph Nodes (normal, abnormal, not done)
- Thyroid (normal, abnormal, not done)
- Musculoskeletal (normal, abnormal, not done)
- Neurological symptoms (normal, abnormal, not done)

### 17.3 Vital Signs

Vital signs will be summarized among adult patients ( $\geq$  18 years at informed consent) by visit. The following vital signs measurements will be reported (see **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported):

- Height (cm)
- Weight (kg)
- Body mass index (BMI) (kg/m<sup>2</sup>)
- Temperature (<sup>0</sup>C)
- Heart Rate (beats/min)
- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy




#### 17.3.1 Derivations

• BMI  $(kg/m^2) = [Weight (kg)/(Height (cm)/100)^2].$ 

### 17.4 Laboratory Evaluations

Clinical laboratory results (hematology, clinical chemistry, urinalysis, and lipid profile) will be summarized (see **Section 8.1** Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported) at each visit.

### 18. EXPLORATORY ANALYSES – EFFECTIVENESS

The exploratory analyses will be performed using the EAS population.

### **18.1** Exploratory Analysis Variables

The exploratory objective is to evaluate the effectiveness achieved with daily SC metreleptin treatment in patients with congenital or acquired generalized lipodystrophy. The exploratory effectiveness variables are:

- hemoglobin A1c (HbA1c)
- fasting plasma glucose
- triglycerides
- leptin/metreleptin concentration

#### 18.2 Exploratory Analysis Description, Derivations, and Definitions

Exploratory variables will be summarized using descriptive statistics (see **Section 8.1** Statistical Summaries, Tests and Confidence Intervals) and results will be presented as described below below:

- by visit
- as absolute change from baseline and percent change from baseline at each visit

HbA1c, fasting plasma glucose, and triglycerides will also be summarized by clinically relevant categories at each visit:

- $\circ$  hbA1c (<8%, >=8%)
- o fasting plasma glucose (<70 mg/dL, >=70 mg/dL and <=100 mg/dL, <100 mg/dL)

| Document: | Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the | | |
|---|---|---|---|
| | Immunogenicity of Daily SC Metreleptin Treatment in Patients with | Generalized Lipodystrophy | |
| | | Version Date: | 131// 1202/ |



o triglycerides (<500 mg/dl, >=500 mg/dl).

See Section 8.1 Statistical Summaries, Tests and Confidence Intervals for a description of statistics to be reported.

#### 19. APPENDIX 1. PARTIAL DATE CONVENTIONS

As applicable, partial dates may be imputed for the purposes of categorizing medications as prior/concomitant and defining TEAs. Imputed dates will NOT be presented in listings. Conventions for imputing partial dates are described below. In general, partial date conventions are designed such that:

- If it is unclear whether or not a medication is prior or concomitant due to partial dates, the worst case will be assumed (i.e., concomitant).
- If it is unclear whether or not an AE is a TEAE due to partial dates, the worst case will be assumed (i.e., TEAE).

If a single medication or AE is reported more than once and partial date imputations cause the instances to appear overlapping, then the medication or AE will be assumed to be a single continuous instance. Start date will be assumed to be the earliest occurring started date (imputed or observed), and end date will be assumed to be the last occurring end date (imputed or observed).

**Table 1: Algorithm for Imputing Partial Dates** 

| Missing data element | | | | Imputation rule |
|---|---|---|---|---|
| Start date or stope date? | Day | Month | Year | |
| Start Date | Yes | No | No | If the non-missing month is the same as the month of study medication start, impute study medication start date. Otherwise, impute the first day of the non-missing month. |
| Start Date | Yes | Yes | No | If the non-missing year is the same as the year of study medication start, impute study medication start date. Otherwise, impute the first day of the non-missing year (i.e., January 1 <sup>st</sup> ). |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


Version Date: 13MAR2024

Copyright © 2018 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



| Start Date | Yes | Yes | Yes | Impute study medication start date. |
|---|---|---|---|---|
| Stop Date | Yes | No | No | If study discontinuation date occurred during the non-missing month, impute study discontinuation date. |
| | | | | Otherwise, impute the last day of the non-missing month. |
| | | | | If study discontinuation date occurred during the non-missing year, impute study discontinuation date. |
| Stop Date | Yes | Yes | No | |
| | | | | Otherwise, impute the last day of the non-missing year (i.e., |
| | | | | December 31 <sup>st</sup> ). |
| Stop Date | Yes | Yes | Yes | Impute study discontinuation date. |

#### 20. APPENDIX 2. WINDOWING CONVENTIONS

The below windowing conventions will be used to categorize all study assessments, including assessments occurring during unscheduled visits, into time periods of interest. Days are counted from the date of baseline visit where Baseline is defined as Day 0.

Only one assessment of each type will be presented from each analysis window. If more than one assessment of the same type occurs within an analysis window, then the maximum severity result will be selected for presentation. If more than one assessment of each types occurs within the maximum severity category, the result closest to the end of the analysis window will be selected. If the concept does not apply, then the result closest to the end of the analysis window will be selected.

The result closest to the end of the analysis window is preferred since the end of the analysis window aligns with the end of the visit window in all cases while the beginning of the analysis window may precede the beginning of the visit window. Therefore, the result closest to the end of the analysis window is most likely to be within the visit window.

**Table 2: Windowing conventions** 

| Study Visit | Study Month | Protocol Specified Visit Window | Analysis Window |
|---|---|---|---|
| Visit 1 (Screening) | Month -1 | Day -28 to Day 0 | Day ≤ -1 |
| Visit 2 (Baseline) | Month 0 | Day 0 | Day 0 |
| Visit 3 | Month 1 | Day 23 to Day 37 | Day 1 to Day 37 |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy





#### Statistical Analysis Plan

| Study Visit | Study Month | <b>Protocol Specified Visit Window</b> | Analysis Window |
|---|---|---|---|
| Visit 4 | Month 2 | Day 53 to Day 67 | Day 38 to Day 67 |
| Visit 5 | Month 4 | Day 114 to Day 128 | Day 68 to Day 128 |
| Visit 6 | Month 6 | Day 175 to Day 189 | Day 129 to Day 189 |
| Visit 7 | Month 9 | Day 266 to Day 280 | Day 190 to Day 280 |
| Visit 8 | Month 12 | Day 350 to Day 378 | Day 281 to Day 378 |
| Visit 9 | Month 18 | Day 533 to Day 561 | Day 379 to Day 561 |
| Visit 10 | Month 24 | Day 715 to Day 743 | Day 562 to Day 743 |
| Visit 11 | Month 30 | Day 898 to Day 926 | Day 744 to Day 926 |
| Visit 12 | Month 36 | Day 1080 to Day 1108 | Day ≥ 927 |

Document: Statistical Analysis Plan: AEGR-734-401: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the

Immunogenicity of Daily SC Metreleptin Treatment in Patients with Generalized Lipodystrophy


**Certificate Of Completion** 

Envelope Id: 32D0AF19B56F4854BFE09C4CF3764A19

Subject: Complete with DocuSign: SAP\_V2.1\_PMR\_DYA76668\_13Mar2024\_CLEAN.pdf

Source Envelope:

Document Pages: 25 Certificate Pages: 5 AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC+09:00) Osaka, Sapporo, Tokyo

Status: Completed

Envelope Originator: Leonor Rodrigues

1 IMS Drive

Plymouth Meeting, 19462 leonor.rodrigues@igvia.com IP Address: 185.76.228.249

**Record Tracking** 

Status: Original

3/14/2024 5:54:11 AM

Holder: Leonor Rodrigues

leonor.rodrigues@iqvia.com

Location: DocuSign

**Signer Events** 

Brian Mangal

b.mangal.consultant@chiesi.com

Security Level: Email, Account Authentication

(None)

Signature DocuSigned by:

Signatures: 4

Initials: 0

Brian Mangal FA68091E7FAE42C

Signature Adoption: Pre-selected Style Using IP Address: 66.183.205.188

**Timestamp** 

Sent: 3/14/2024 6:02:58 AM Resent: 3/19/2024 12:41:11 AM Viewed: 3/20/2024 6:52:33 AM Signed: 3/20/2024 6:52:46 AM

**Electronic Record and Signature Disclosure:** 

Accepted: 3/20/2024 6:52:33 AM ID: a060b1a1-2451-4018-8df2-c5701de3cbb5

Company Name: IQVIA

Imaani Easthausen

imaani.easthausen@igvia.com

Security Level: Email, Account Authentication

(None)

Imaani Easthausen

C8854A1FE2E8486...

DocuSigned by:

Signature Adoption: Pre-selected Style Using IP Address: 162.44.245.32

Sent: 3/14/2024 6:02:59 AM Viewed: 3/14/2024 6:03:48 AM Signed: 3/14/2024 6:03:54 AM

**Electronic Record and Signature Disclosure:** 

Accepted: 7/5/2023 10:40:01 PM

ID: 6a3dec7a-0b89-4130-9ad3-99dfd386f4f5

Company Name: IQVIA

Janet Boylan

janet.boylan@chiesi.com

Security Level: Email, Account Authentication

(None)

DocuSigned by: Janet Boylan

Signature Adoption: Pre-selected Style Using IP Address: 78.152.221.250

Sent: 3/14/2024 6:02:59 AM

Resent: 3/19/2024 12:41:12 AM Viewed: 3/28/2024 3:36:15 AM

**Electronic Record and Signature Disclosure:** 

Accepted: 3/28/2024 3:36:15 AM

ID: 400f6e02-f0ce-43f3-93b7-743217482d53

Company Name: IQVIA

Orla Casey

orla.casey@chiesi.com

Security Level: Email, Account Authentication

(None)

Oda Casey 957F4F8B479F407

Signature Adoption: Pre-selected Style

Signed: 3/28/2024 3:36:28 AM

Sent: 3/14/2024 6:03:00 AM Resent: 3/19/2024 12:41:12 AM Viewed: 3/19/2024 10:58:15 PM Signed: 3/19/2024 10:59:13 PM

Using IP Address: 37.228.226.45

**Electronic Record and Signature Disclosure:** 

| Accepted: 2/12/2024 5:02:33 AM ID: ca06339e-3781-458b-99d1-cfe2c26a3dab Company Name: IQVIA | | |
|---|---|---|
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 3/14/2024 6:03:00 AM<br>3/19/2024 10:58:15 PM<br>3/19/2024 10:59:13 PM<br>3/28/2024 3:36:28 AM |
| Payment Events | Status | Timestamps |

Timestamp

Signature

Signer Events

**Electronic Record and Signature Disclosure** 

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

## Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

## **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### **How to contact IOVIA:**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

## 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

## 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

## 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

## Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.




Client: Chiesi

 Protocol No.:
 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

### The timing of the change(s) was:

After authorization (signed version) of the SAP but prior to the database lock/interim data cut/ final Statistical Report/ Clinical Study Report (CSR)

After database lock/ interim data cut/ final Statistical Report/ CSR

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

Describe the change(s) required:

Form No: RWI\_FM\_BIOS0027 Revision 2 Reference: RWI\_WI\_BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

### Changes documented in 16Dec2024 version (prior to DBL)

1. Update definition of EAS from:

[E]nrolled subjects who received at least one documented dose of metreleptin and who have baseline and post-dose laboratory results on the measure of interest at the time point of interest.

To:

Enrolled subjects who received at least one documented dose of metreleptin and who have at least one anti-metreleptin/anti-HuL binding antibody (Antidrug Antibody (ADA) binding) result.

2. Update the following analysis from:

AEs, serious AEs (SAEs), AEs of special interest (AESIs), TEAEs, AEs possibly caused by metreleptin, and AEs leading to metreleptin discontinuation will be summarized by ADA positivity and titer, cell-based NAb positivity and titer, and RB positivity, titer, and quintile of percent inhibition.

To:

TEAEs, serious TEAEs, TEAEs that are AEs of special interest (AESIs), TEAEs possibly caused by metreleptin, and TEAEs leading to metreleptin discontinuation will be summarized by ADA positivity and titer, cell-based NAb positivity and titer, and RB positivity, titer, and quintile of percent inhibition.

3. Update analysis windows such that data collected for a CRF-defined visit are windowed according to the CRF-defined visit. Previously analysis windows ended on the same day as CRF-defined visit windows and extended CRF-defined windows to cover the calendar space since the last CRF-defined visit. Analysis windows are updated to extend CRF-defined visit windows to cover calendar space on either side of the CRF-defined visit window. See updated windows in Table 1 below.

## Changes added 26Feb2025 (after DBL)

4. Treatment interruptions occurred for Patient 002002 from 07-Jun-2021 to 01-Jul-2021 and Patient 002003 from 22-Feb-2021 to 27-Feb-2021. These treatment interruptions were not recorded in the "Prescription Changes to Metreleptin" CRF, but were confirmed by the site investigator. These prescription changes will be hard coded. Request made by: Chiesi. Date of request: 21-Feb-2025.

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

### **Datasets/programs Impacted:**

Dataset: EXProgram: EX.sas

- Program details: For subject "002002" create extra rows for temporary drug interruption where start date is "2021-06-07" and end date is "2021-07-01". Also, for subject "002003" create extra rows for temporary drug interruption where start date is "2021-02-22" and end date is "2021-02-27". The EXCAT for these new rows will be "PRESCRIPTION CHANGES TO METRELEPTIN". Set EXDOSE equals to 0 mg and for temporary interruption questionnaire (Did the prescription change result in a temporary interruption of treatment?) equals to "Yes".
- Program log notes: NH02/24/2025 : Create treatment interruption rows for Patient 002002 from 07-Jun-2021 to 01-Jul-2021 and Patient 002003 from 22-Feb-2021 to 27-Feb-2021 as confirmed by the site investigator under RSC dataset i.e. Prescription Changes to Metreleptin.
- Implementer: Narek Hovhannisyan
- QC Programmer: Anita Panthi

#### TLFs Impacted:

- Table 1.6 Metreleptin exposure (SAF)
  - Any temporary interruptions and number of temporary interruptions
  - Any dose reductions
  - Duration of exposure accounting for interruptions (months)
- Listing 12 Prescription changes to metreleptin (SAF)
- Figure 6.2 Patient 002002 Profile: Immunogenicity and effectiveness
- Figure 6.3 Patient 002003 Profile: Immunogenicity and effectiveness

#### Impact on Interpretation of results:

Improves interpretability of results as confirmed data not included in database are presented in analyses.

5. Patients 002003 and 004004 had inconsistent results in RB samples at Visit 5 (Month 4) and Visit 4 (Month 2), respectively. Specifically, testing at the minimum required dilution (dilution factor = 6) with acid was positive at Tier 1 (initial test), but negative at Tier 2 (re-test). Given inconsistent results, these samples were

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

removed from summary analyses using hard coding. Request made by: Chiesi. Date of request: 10-Jan-2025.

#### **Datasets/programs Impacted:**

- Dataset: ADIS
- Program: ADIS.sas
- Program details: If Subject '002003' and AVISIT is 'Month 4' then keep ANL02FL blank, In addition, if Subject '004004' and AVISIT is 'Month 2', then keep ANL02FL blank.
- Program log notes: [notes] AP:2/11/2025 Update usubjid = 'AEGR-734-401-002003' and avisit = 'Month 4' and usubjid = 'AEGR-734-401-004004' and avisit = 'Month 2' analysis results as NOT REPORTABLE s these are inconsistent results as confirmed by sponsor.
- Implementer: Anita Panthi
- QC Programmer: Nicolas Dalcero

#### TLFs Impacted:

- Table 4.1 RB activity at MRD among ADA positive patients (EAS)
  - RB positivity by time point
- Table 4.2 RB activity by titer among ADA positive patients (EAS)
  - o RB titer by time point
- Table 4.3 RB percent inhibition at MRD among RB positive patients (EAS)
  - RB percent inhibition at MRD by time point
- Table 4.4 Ever RB positive and peak RB activity among ADA positive patients (EAS)
  - Time to RB positivity
  - Time to peak RB
- Figure 1.3 RB activity by patient among ever ADA positive patients (EAS)
  - o RB titer by timepoint
- Figure 6.3 Patient 002003 Profile: Immunogenicity and effectiveness
  - RB titer by timepoint
- Figure 6.9 Patient 004004 Profile: Immunogenicity and effectiveness
  - RB titer by timepoint

#### Impact on Interpretation of results:

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

Improves interpretability, because uninterpretable results are removed from summary analyses.

6. For patients 004004 and 004005, ADA samples were tested beyond the recommended number of freeze/thaw cycles. Re-analysis of aliquots with lower number of freeze/thaw cycles was possible, and study team agreed that the retested samples should be included in summary tables. As the algorithm used to select ADA results for inclusion in summary tables was already selecting the retested samples for inclusion in summary tables, no modifications were required. Request made by: Chiesi. Date of request: 11-Mar-2025.

Datasets/programs Impacted: None.

TLFs Impacted: None.

**Impact on Interpretation of results:** No changes.

 Treatment interruption for Patient 003001 was not recorded in Prescription Change Log, but was identified in AEs where action taken with metreleptin was recorded as "drug interrupted." Treatment interruption start and end dates were imputed as start date of pregnancy (18-Jun-2020, AE ID: 1) and end date of miscarriage (23-Jul-2020, AE ID: 3).

#### **Datasets/programs Impacted:**

Dataset: ADEX

Program: ADEX.sas

Program details: For subject "003001" - create extra rows for temporary drug interruption where start date is "2020-06-18" and end date is "2020-07-23". The EXCAT for these new rows will be "PRESCRIPTION CHANGES TO METRELEPTIN". Set EXDOSE equals to 0 mg and for temporary interruption questionnaire (Did the prescription change result in a temporary interruption of treatment?) equals to "Yes".Program log notes: BN03/20/2025 : Create treatment interruption rows

notes: BN03/20/2025 : Create treatment interruption rows for Patient 003001 from 18-Jun-2020 to 23-Jul-2020 as confirmed by the site investigator under PRSC dataset i.e. Prescription Changes to Metreleptin.

Reference: RWI WI BIOS0015

Implementer: Barbara NogarQC Programmer: Anita Panthi

Form No: RWI\_FM\_BIOS0027 Revision 2




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

### **TLFs Impacted:**

- Table 1.6 Metreleptin exposure (SAF)
  - Any temporary interruptions and number of temporary interruptions
  - Any dose reductions
  - Duration of exposure accounting for interruptions (months)
- Listing 12 Prescription changes to metreleptin (SAF)
- Figure 6.2 Patient 002002 Profile: Immunogenicity and effectiveness
- Figure 6.3 Patient 002003 Profile: Immunogenicity and effectiveness

### Impact on Interpretation of results:

Improves interpretability of results as data not included in database are presented in analyses.

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

### **Table 1: Updated Visit Windows**

| Study Visit | Study Month | Protocol Specified Visit Window | Analysis Window |
|---|---|---|---|
| Visit 1 (Screening) | Month -1 | Day -28 to Day 0 | Day ≤ -1 |
| Visit 2 (Baseline) | Month 0 | Day 0 | Day 0 |
| Visit 3 | Month 1 | Day 23 to Day 37 | Day 1 to Day 44 |
| Visit 4 | Month 2 | Day 53 to Day 67 | Day 45 to Day 90 |
| Visit 5 | Month 4 | Day 114 to Day 128 | Day 91 to Day 151 |
| Visit 6 | Month 6 | Day 175 to Day 189 | Day 152 to Day 227 |
| Visit 7 | Month 9 | Day 266 to Day 280 | Day 228 to Day 314 |
| Visit 8 | Month 12 | Day 350 to Day 378 | Day 315 to Day 455 |
| Visit 9 | Month 18 | Day 533 to Day 561 | Day 456 to Day 637 |
| Visit 10 | Month 24 | Day 715 to Day 743 | Day 638 to Day 820 |
| Visit 11 | Month 30 | Day 898 to Day 926 | Day 821 to Day 1002 |
| Visit 12 | Month 36 | Day 1080 to Day 1108 | Day ≥ 1003 |

Describe the process used to decide on the change(s) and who was involved:

## Changes documented in 16Dec2024 version (prior to DBL)

Discussed with client at meetings on 11Sep2024 and 14Oct2024.

### Changes added 26Feb2025 (after DBL)

Discussed with client via email and at meetings on 06Feb2025 and 07Feb2025.

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

 AEGR-734-401

 Project Code:
 DYA76668

 Date:
 26-Feb-2025

The group(s) responsible for the change(s) and implications for the study:

### Changes documented in 16Dec2024 version (prior to DBL)

Imaani Easthausen – Statistical Team Lead, IQVIA

Petya Angelova – Medical Lead, IQVIA

Orla Casey - Translational and Immunogenicity, Chiesi

Janet Boylan – Head of Clinical Operations Chiesi

Inbar Aviezer- Associate Clinical Project Manager, Chiesi

Meng Wang – Statistician, Chiesi

Sue Schmidt - Consultant Immunogenicity Subject Matter Expert, Chiesi

Roberto Pierini – Immunogenicity Subject Matter Expert, Chiesi

Brian Mangal - Consultant Statistician, Chiesi

### Changes added 26Feb2025 (after DBL)

Imaani Easthausen – Statistical Team Lead, IQVIA

Orla Casey - Translational and Immunogenicity, Chiesi

Janet Boylan – Head of Clinical Operations Chiesi

Inbar Aviezer- Associate Clinical Project Manager, Chiesi

Meng Wang – Statistician, Chiesi

Roberto Pierini – Immunogenicity Subject Matter Expert, Chiesi

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015




Client: Chiesi

Protocol No.: AEGR-734-401
Project Code: DYA76668

Date: 26-Feb-2025

Form completed by:

Title Name Signature Date

Statistical Team Imaani Easthausen

Lead Imaani Easthausen 15-Apr-2025

Form approved by:

Title/ Role Name Signature Date

Senior Tracy Franklin — Docusigned by:

Biostatistical
Reviewer 15-Apr-2025

Form approved by:

Title Name Signature Date

DocuSigned b

Lead Shahrzad Salmasi Shahrzad Salmasi 15-Apr-2025

Form approved by Client Representative (if applicable):

Title Name Signature Date

Translational and Orla Casey

Immunogenicity
Lead

Docusigned by:

24-Apr-2025

<del>957E4F0B479F407...</del>

Head of Clinical Janet Boylan
Operations

Janet Boylan 23-Apr-2025

Form No: RWI FM BIOS0027 Revision 2 Reference: RWI WI BIOS0015



#### **Certificate Of Completion**

Status: Completed Envelope Id: 35BA08F0-967F-4C52-BCC8-53059503E4E4

Subject: Complete with Docusign: Changes to Planned Analyses\_SAP\_V2.1\_PMR\_DYA76668\_01Apr2025.docx

Source Envelope:

Document Pages: 10 Signatures: 5 Envelope Originator: Initials: 0 Imaani Easthausen Certificate Pages: 5 AutoNav: Enabled 1 IMS Drive

Envelopeld Stamping: Enabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Plymouth Meeting, 19462 imaani.easthausen@iqvia.com IP Address: 162.44.245.32

#### **Record Tracking**

Status: Original Holder: Imaani Easthausen Location: DocuSign

4/15/2025 9:23:50 AM imaani.easthausen@iqvia.com

### **Signer Events**

Signature Imaani Easthausen

Security Level: Email, Account Authentication

(None)

DocuSigned by: Imaani Easthausen C8854A1FE2E8486..

Signature Adoption: Pre-selected Style Using IP Address: 162.44.245.32

### **Timestamp**

Sent: 4/15/2025 9:26:43 AM Viewed: 4/15/2025 9:26:51 AM Signed: 4/15/2025 9:27:01 AM

#### **Electronic Record and Signature Disclosure:**

Accepted: 7/5/2023 9:40:01 AM ID: 6a3dec7a-0b89-4130-9ad3-99dfd386f4f5

Company Name: IQVIA

imaani.easthausen@iqvia.com

Janet Boylan

janet.boylan@chiesi.com

Security Level: Email, Account Authentication

(None)

DocuSigned by Janet Boylan A5E2C5EA84644FC

Signature Adoption: Pre-selected Style Using IP Address: 144.2.246.98

### Sent: 4/15/2025 9:26:44 AM Viewed: 4/23/2025 6:23:36 AM Signed: 4/23/2025 6:24:13 AM

#### **Electronic Record and Signature Disclosure:**

Accepted: 3/27/2024 2:36:15 PM

ID: 400f6e02-f0ce-43f3-93b7-743217482d53

Company Name: IQVIA

Orla Casey

orla.casey@chiesi.com

Security Level: Email, Account Authentication

(None)

DocuSigned by: Orla Casey 957E4F8B479F407.

Signature Adoption: Pre-selected Style Using IP Address: 64.43.50.97

Sent: 4/15/2025 9:26:44 AM Viewed: 4/24/2025 10:18:23 AM Signed: 4/24/2025 10:55:17 AM

#### **Electronic Record and Signature Disclosure:**

Accepted: 2/11/2024 3:02:33 PM

ID: ca06339e-3781-458b-99d1-cfe2c26a3dab

Company Name: IQVIA

Shahrzad Salmasi

shahrzad.salmasi@iqvia.com

Security Level: Email, Account Authentication

(None)

Shalirzad Salmasi

Signature Adoption: Pre-selected Style Using IP Address: 162.44.245.32

Sent: 4/15/2025 9:26:44 AM Viewed: 4/15/2025 5:48:11 PM Signed: 4/15/2025 5:48:25 PM

#### **Electronic Record and Signature Disclosure:**

**Signer Events** 

**Signature** 

**Timestamp** 

Accepted: 4/15/2025 5:48:11 PM ID: 05bf8adc-adb8-406d-b320-096bb65cf5c2

Company Name: IQVIA

Tracy Franklin

Tracy.Franklin@quintiles.com

Tracy Franklin

Security Level: Email, Account Authentication

(None)

Tracy Franklin

Signature Adoption: Pre-selected Style Using IP Address: 162.44.245.32

Sent: 4/15/2025 9:26:44 AM Viewed: 4/15/2025 12:14:22 PM Signed: 4/15/2025 12:14:29 PM

### **Electronic Record and Signature Disclosure:**

Not Offered via Docusign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 4/15/2025 9:26:44 AM<br>4/15/2025 12:14:22 PM<br>4/15/2025 12:14:29 PM<br>4/24/2025 10:55:17 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

## **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### **How to contact IOVIA:**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

## 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

## 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

## 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

## Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.